CLINICAL TRIAL: NCT01789333
Title: Study of the Safety and Effectiveness of Photochemically Induced Collagen Cross- Linking at Higher Irradiances in Patients With Keratoconus or Ectasia
Brief Title: Higher Irradiance in Keratoconus Ectasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Trokel (Other)
Responsible Party: Sponsor-Investigator, Stephen Trokel, Professor of Clinical Ophthalmology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF4157
Record Dates: First submitted 2012-11-20; First posted 2013-02-12 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus; Ectasia
Keywords: Keratoconus; Ectasia; UVA light; riboflavin; post-LASIK; irregular astigmatism
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Riboflavin; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: 30 patients will be treated at 9 mw/cm2.
Oversight: Data Monitoring Committee: No

ARMS (1):
- 9 mw/cm2 at 10 minutes group (Experimental): 30 patients will be treated with UVA light source at 9 mw/cm2 at 10 minutes. Drug: Riboflavin Dose:1 drop every 2 to 3 minutes for 15 to 20 minutes
  Interventions: Device: UVA Light with irradiance exposure of 9 mW/cm2; Drug: Riboflavin 0.1% ophthalmic solution

INTERVENTIONS:
Device: UVA Light with irradiance exposure of 9 mW/cm2 — The device's light emitting diode (LED) is used to deliver a metered dose of Ultraviolet A (UVA) light to a targeted treatment area for illuminating the cornea during corneal collagen cross-linking.
  The aperture setting will be set at 10 mm, and the eye will be irradiated for 10 minutes for the high irradiance exposure of 9 milliwatts (mW)/cm2. During the exposure, instillation of riboflavin will continue (1 drop every 3 minutes).
Drug: Riboflavin 0.1% ophthalmic solution — The speculum is removed and one (1) drop of Riboflavin 0.1% ophthalmic solution will be instilled topically in the eye every 3 minutes for 30 minutes. At the end of the 30 minute riboflavin pre-treatment period, the eye will be examined to assure the presence of a yellow flare in the anterior chamber, indicating riboflavin saturation of the corneal tissue. If the yellow flare is not detected, riboflavin will continue to be instilled until the presence of the yellow flare in the anterior chamber is confirmed.
  During UVA irradiation, instillation of riboflavin will be continued every 3 minutes. For a 30-minute pre-treatment and 30-minute irradiation, the total dose of riboflavin solution is approximately 32 drops, or 1.6 ml (1 drop = 0.05 ml; 1.6 mL = 1.6 mg riboflavin).
  Other Names: Riboflavin

SUMMARY:
The purpose of the study is to see if brighter lights will allow for shortening of the treatment time required to stabilize the eyes of patients with keratoconus or a bulging cornea. The investigators will be comparing the therapeutic effects of two different higher brightnesses of ultra violet light on a riboflavin treated eye. One light will be twice as bright as the other and the exposure time of these brighter lights to deliver equivalent energy to the cornea will be reduced from the standard 30 minutes to 10 and 5 minutes. Riboflavin is vitamin B2 and the investigators are trying to determine if an identical clinical effect can be achieved the brighter treatment lights are used for shorter times. The investigators will also monitor the clinical effect and the status of the cornea to see if additional risks are associated with the brighter light.

ELIGIBILITY:
Inclusion Criteria:

Subjects who have one or both eyes that meet two of the following criteria will be considered candidates for this study:

1. 16 years of age or older
2. Having a diagnosis of progressive keratoconus or pellucid marginal degeneration.

   1. Characteristic pattern of deformity as analyzed by the Pentacam map.
   2. Minimal thickness of 350 microns
3. The ability to sign a written informed consent
4. States a willingness and ability to comply with schedule for follow-up visits
5. Subject willing to remove contact lenses prior to evaluation and treatment

Inclusion criteria for ectasia

1. History of having undergone a keratorefractive procedure and show:

   1. Steepening by Pentacam study
   2. Thinning of cornea
   3. Shift in the position of thinnest portion of cornea
   4. Unstable refraction with increasing myopia and astigmatism
   5. Development of irregular astigmatism
2. At least two of the above criteria must be present.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from this study:

Subjects meeting any of the following criteria will be excluded from this protocol:

1. Eyes classified as either normal or atypical normal,
2. Corneal pachymetry ≤ 350 microns at the thinnest point in treatment zone measured by Pentacam.
3. A history of delayed epithelial healing.
4. Pregnancy (including plan to become pregnant) or lactation during the course of the study
5. A known sensitivity to study medications
6. Patients with nystagmus or any other condition that is severe enough to prevent steady gaze during the treatment
7. Inability to cooperate with diagnostic tests.
8. Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.
9. Patients who are unable to remain supine and tolerate a lid speculum.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Total Optical Aberrations of the Cornea following Cross-Linking | Baseline to 6 months
  Assessment of changes in corneal curvature, as analyzed using a Pentacam Scheimpflug Analyzer will be used in all patients. This allows measurement of corneal thickness, maximum and minimum curvatures and aberration analysis of the cornea as an optical element. The most significant objective measure of change is the total Higher Order Aberrations of the cornea and the Kmax, or steepest curvature of the cornea. Analysis of corneal curvature is directly related to improvement in the corneal shape which is directly related to visual function.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Trokel, MD, Principal Investigator — Columbia University
Locations (1):
- Edward Harkness Eye Institute-Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided